CLINICAL TRIAL: NCT01294254
Title: Open, Prospective, Controlled, Randomised, Multicenter Phase II Clinical Trial to Compare Intra-individually the Efficacy and Tolerance of Oleogel-S10 Versus Moist Wound Healing Dressing Alone in Accelerating the Epithelialization of Split Thickness Skin Graft Donor Sites
Brief Title: Trial to Compare Intra-individually the Efficacy and Tolerance of Oleogel-S10 Versus Moist Wound Healing Dressing Alone in Accelerating the Epithelialization of Split Thickness Skin Graft Donor Sites
Acronym: OleoSplit
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Birken AG (Industry)
Responsible Party: Sponsor
Organization: Amryt Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSH-10
Record Dates: First submitted 2010-04-14; First posted 2011-02-11 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Accelerating the Epithelialization of Split Thickness Skin Graft
Keywords: wound reepithelialization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimantal: wound site will be treated with Oleogel-S10 (Experimental): The patients will be randomised in a ratio of 1:1 with regard to the part of the skin graft donor site that is treated with Oleogel-S10.
  Arm A: application of Oleogel-S10 towards the periphery of the body, i.e. the lower part of the leg
  Arm B: application of Oleogel-S10 towards the centre part of the body, i.e. the upper part of the leg
  * Oleogel-S10 on one half of the skin graft donor site (each time when the wound dressing is changed during a time period of 14 days, normally once daily)
  * Moist wound healing dressings alone (Mepilex) on the other half of the skin graft donor site
  Interventions: Drug: Oleogel-S10
- Moist wound healing dressing alone (Active Comparator): Treatment with moist wound healing dressings alone (Mepilex) on the other half of the skin graft donor site
  Interventions: Procedure: Moist wound healing dressings alone (Mepilex) on the other half of the skin graft donor site

INTERVENTIONS:
Drug: Oleogel-S10 — Oleogel-S10 on one half of the skin graft donor site (each time when the wound dressing is changed during a time period of 14 days, normally once daily)
  Arms: experimantal: wound site will be treated with Oleogel-S10
Procedure: Moist wound healing dressings alone (Mepilex) on the other half of the skin graft donor site — wound is covered conventionally by applying one half of the Mepilex cut
  Arms: Moist wound healing dressing alone

SUMMARY:
In this study the wound reepithelialization of that part of the skin graft donor site, which is treated with Oleogel-S10 compared to that part of the wound, which is covered by moist wound healing dressing alone will be investigated.

DETAILED DESCRIPTION:
As a first step, an adequate size of the wound healing dressing (Mepilex) is taken and cut in half. Then, half of the SSG (split skin graft) wound is covered conventionally by applying one half of the Mepilex cut. Afterwards Oleogel-S10 is applied to the other half of the Mepilex cut, which is used to cover the other half of the SSG wound. Both parts of the Mepilex dressings are then covered by an additional conventional dressing.

Oleogel-S10 is always applied to the same part of the SSG wound for each patient, respectively, depending on the randomization of the patient, either towards the periphery of the body, i.e. the lower part of the leg, or towards the centre part of the body, i.e. the upper part of the leg. In order to avoid a confusion about which part has to be treated with Oleogel-S10, the healthy skin next to the SSG wound will be marked with ink for indication of the Oleogel-treated part of the wound.

Each day during the treatment period, whenever the wound dressing is changed, a clinical examination and assessment of the progress of epithelialization of the SSG wound will be conducted, including evaluation of tolerance, and photos of the wound without dressing will be taken.

A blinded assessment of the efficacy is conducted by two independent investigators using the macro-photos of every day, when wound dressings were changed, and a final examination is done. In this assessment, the third part of the SSG wound that is in between the left and right parts is neglected.

ELIGIBILITY:
Inclusion Criteria:

Patients may participate in the study if they have/are

* Patients aged 18-95 years who have provided written informed consent.
* Patients requiring skin grafting due to burns, trauma, chronic venous ulcers, or surgical removal of cutaneous malignancies with a donor site expected to be between 8 and 200 cm2 on a non-articulated area.
* Patient is prepared to comply with all study requirements, including the following:

  * Application of Oleogel-S10 on the SSG at every change of wound dressing;
  * Regular clinic visits during the treatment period, and follow-up period.
* Negative pregnancy test of women of childbearing potential performed within 7 days prior to the start of treatment.
* Women of childbearing potential must agree to use an effective method of contraception (Pearl-Index < 1, e.g. hormonal contraception including the combined oral contraceptive pill, the transdermal patch, and the contraceptive vaginal ring, intrauterine devices or sterilization) during treatment and for at least 6 months thereafter.
* Men must agree to use an effective method of contraception during treatment and for at least 6 months thereafter.

Exclusion Criteria:

Patients will be excluded from the study if they have/are

* burns involving more than 15% of their total body area;
* sepsis, haemodynamic instability requiring pressor support or positive blood microbiology cultures within 48h of surgery;
* inhalation injury requiring artificial respiratory assistance;
* requiring skin grafts following removal of suspicious skin lesions;
* received treatment with systemic steroids during the 30 days prior to surgery;
* uncontrolled diabetes or diabetic ulcers;
* diseases or conditions that could, in the opinion of the Investigator, interfere with the assessment of safety, tolerance or efficacy;
* previously skin grafts harvested from the area to be studied;
* a skin disorder that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial;
* a history of clinically significant hypersensitivity to any of the drugs or surgical dressings to be used in this trial;
* known multiple allergic disorders;
* taking, or have taken, any investigational drugs within 3 months prior to the screening visit;
* undergoing investigations or changes in management for an existing medical condition;
* not likely to complete the trial for whatever reason.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Wound reepithelialization of that part of the skin graft donor site, which is treated with Oleogel-S10 compared to that part of the wound, which is covered by moist wound healing dressing alone during a treatment period of 14 days. | 14 days

SECONDARY OUTCOMES:
• Size of wound epithelialization | 3 months
• Touch sensitivity: Sensitivity of the SSG wound by touching it with a spatula or cotton swabs (visual analogue scale from "no" = 0 to "severe" = "10" | 3 months
• Pruritus (visual analogue scale from "no" = 0 to "strong" = "10") | 3 months
• Reconstitution of the skin (% reepithelization) 3 months after skin explantation | 3 months
  Evaluation of wound closure by assessment of epithelialization (in %)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Robert Metelmann, Prof. Dr. med., Principal Investigator — University Hospital of Ernst-Moritz-Arndt-University Greifswald
Locations (2):
- Germany (2):
  - Universitäts-Hautklinik Freiburg, Freiburg im Breisgau
  - Universitätsklinikum der Ernst-Moritz-Arndt-Universität Greifswald, Greifswald

REFERENCES:
- [Result] Metelmann HR, Brandner JM, Schumann H, Bross F, Fimmers R, Bottger K, Scheffler A, Podmelle F. Accelerated reepithelialization by triterpenes: proof of concept in the healing of surgical skin lesions. Skin Pharmacol Physiol. 2015;28(1):1-11. doi: 10.1159/000357501. Epub 2014 Jul 15. PMID 25034442